CLINICAL TRIAL: NCT05382949
Title: SilverBills: A Financial and Legal Tech Tool for Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marci Lobel-Esrig (Other)
Responsible Party: Sponsor-Investigator, Marci Lobel-Esrig, CEO and Founder, Silverbills, Inc.
Organization: Silverbills, Inc. (Other)
Other Study IDs: 074126
Record Dates: First submitted 2022-05-06; First posted 2022-05-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Caregiver Burden
Keywords: Financial Management; Well-being; Dementia; Legal Management; Caregiver; Stress
MeSH Terms: conditions — Caregiver Burden; Dementia | interventions — Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SilverBills Financial and Legal Tech Tool for Caregivers — All subjects will be receiving the Silverbills financial and legal tech tool and a pre-post analysis will be conducted.

SUMMARY:
Financial and legal management for persons with dementia (PwD) is a crucial responsibility of caregivers. This responsibility adds to the stress and strain of caregiving. Current technology tools that help with bill management and budgeting often require a high degree of technical expertise and provide an insufficient degree of personal support to address the caregivers' needs. Current approaches to financial management are typically aimed at technologically savvy millennials rather than caregivers. Additionally, these approaches do not address the need for safe and accessible storage of legal documents. Thus, the current solutions available for these tasks are a mismatch for caregivers. The investigators will address the lack of effective financial management and legal support for caregivers of PwD. Using proprietary technology, SilverBills receives, scrutinizes, stores, and pays bills on behalf of clients. The goal of this project is to decrease the stress and strain on caregivers of PwD, by providing a simple, safe, and effective financial and legal management tool. The investigators aim to build an easy to use, customizable, client facing application for caregivers to direct the financial activities of PwD. In addition, The investigators will enhance the capabilities of the application to reconcile banking information, detect fraud, secure data, provide enhanced reporting capabilities and provide further budgeting and planning functionality. Finally, in collaboration with researchers from the University of Denver, The investigators will assess caregiver burden and physical, financial, and emotional distress. The team supporting Silverbills V2 includes expertise in elder law, business development, Ruby on Rails software engineering, financial security and cognitive health, caregiving, research design and statistics. The work proposed should demonstrate that the SilverBills V2 product will: 1) Provide a financial management tool which includes a messaging system and vault of critical documents for caregivers of PwD and/or older adults, and 2) Evaluate the effectiveness of our product to decrease caregiver stress and increase caregiver quality of life. This team will support the rigorous scientific validation which will potentially provide evidence of our innovation and support this critical work to provide technological tools for financial and legal management to caregivers of PwD.

DETAILED DESCRIPTION:
Research has demonstrated that education, information and support improve caregiver wellbeing, improve their mental health, and delay the need to move the persons with dementia (PwD) to along-term care setting. Caregivers are often responsible for managing the legal and financial affairs for PwD. This responsibility adds to the stress and strain of caregiving. The SilverBills client-facing application provides an easy to use, efficient financial and legal management tool to caregivers, decreasing caregiver burden. In order to assess the effectiveness of the SilverBills tool, the investigators will measure caregiver burden as well as mental, physical and financial health (baseline and post-intervention).

Research Questions:

1. What are the effects of a client-facing application on the primary outcome (caregiver burden) between baseline (T1) and end (T2) of the study?
2. What are the effects of a client-facing application on the secondary outcomes (mental, physical, and financial health) between T1 and T2?
3. What are the moderators of the effects of client-facing application on the primary outcome and secondary outcomes between T1 and T2?

To achieve the aims of this proposal, recruited participants will remotely and electronically (via Qualtrics data collection software) provide informed consent for research. Participants will be recruited as detailed in the recruitment and retention plan. Participants will meet the following screening criteria: a) Participants must be caregivers aged 18 or above; b) participants must be caregivers of people with dementia; and c) participants are able to provide consent without the aid of another individual.

Participants will complete two surveys at two different time intervals. The first survey will take place at the outset of the research study when the participants are enrolled (T1). The second and final survey will be administered 6 months after the start of the study (T2). The entirety of the data collected throughout this project will be converted into password-protected files (e.g. xlsx), which will be stored in secured electronic platforms (i.e. password-protected OneDrive) that only select team members will have access to. Survey items will be multiple choice and should take respondents no more than 15-20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Provide care for an individual with Dementia

Exclusion Criteria:

* Age <18
* Lack of cognitive capacity to independently consent and complete participation (i.e., one who would require an informant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit approximately 150 caregivers who provide care for an individual with dementia that meet inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden | 1 year
  Zarit Burden Interview

SECONDARY OUTCOMES:
Mental Health | 1 year
  Anxiety and Depression using PHQ-9 and GAD-7
Physical Health | 1 year
  Physical health component of SF-12
Financial Distress | 1 year
  InCharge Financial Distress/Financial Well-Being Scale. Items are measured on a scale of 1 to 10, wherein 1 signifies significant financial concern and 10 signifies little or no financial concern.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chess, MD/JD, Principal Investigator — University of Denver
Locations (1):
- Silverbills, Inc., New Rochelle, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Knoebel Institute for Healthy Aging - University of Denver — https://ritchieschool.du.edu/aging/participate-support